CLINICAL TRIAL: NCT00908193
Title: Assistance Robotics for the Surgical Treatment of the Abdominal Wall Hernia
Brief Title: Laparoscopic "DA VINCI" Robot Assisted Abdominal Wall Hernia Repair
Acronym: ARTE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P051080
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Abdominal Wall Hernia
Keywords: Treatment of abdominal ruptured; Digestive system disease; Coelioscopy; Assistance robotics; Medical device; DA VINCI Robot; Pain patient; Morphine consumption; Comparative Randomized study; patient over 18 years; with ruptured abdominal; with an indication of treatment of ruptured
MeSH Terms: conditions — Hernia, Abdominal; Digestive System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): robot-assisted coelioscopy
  Interventions: Device: Laparoscopic DA VINCI Robot Assisted coelioscopy
- 2 (Active Comparator): conventional coelioscopy
  Interventions: Procedure: conventional coelioscopy

INTERVENTIONS:
Device: Laparoscopic DA VINCI Robot Assisted coelioscopy — Patients with abdominal wall hernia will be treated by robot-assisted coelioscopy for the poses of abdominal plate
  Other Names: Laparoscopic DA VINCI Robot Assisted abdominal coelioscopy
  Arms: 1
Procedure: conventional coelioscopy — Patients with abdominal wall hernia will be treated by conventional coelioscopy for the poses of abdominal plate
  Arms: 2

SUMMARY:
The aim of this study is to prove the superiority of the robotic assistance in laparoscopic repair of abdominal wall hernias .

In this monocentric randomized controlled trial, the use of the DA VINCI robot might reduce the post-operative pain of the patient resulting in a 40% reduction of morphine consumption.

DETAILED DESCRIPTION:
Laparoscopic Robot Assisted abdominal wall hernia repair : a prospective randomized trial:

The main judgement criterion is post operative pain reflected by morphine consumption during the first 48 hours. Secondary criteria are morbidity, quality of life, duration of surgery, conversion rate, complications, the the length of stay and hospital costs.

In this single centre study, inclusion criteria are age above 18, no previous repair of the hernia with a mesh and a diameter of the parietal defect of less than 10 cm. Contraindications are chronic use of pain drugs of level II or above and renal insufficiency (clearance <30ml/min).

The robotic repair was described in a previous paper of our group and will be compared to our classical laparoscopic repair technique, and in both cases with the use of the same prosthetic mesh.

A total of 70 patients to be included in an 18 months period was calculated to prove a 40% reduction in morphine consumption during the postoperative 48h (α=5% and β=10%).

The total duration of the study is 30 months (12 months of follow-up for each patient).

ELIGIBILITY:
Inclusion Criteria:

* over 18 years
* with indication of hernia repair
* a collar with a diameter of less than 10cm
* no antecedent of hernia treatment with poses plate
* agreeing coelioscopy
* agreeing to participate the clinical study, having sign an informed consent
* agreeing a regular monitor

Exclusion Criteria:

* taking analgesic tier 2 or 3
* against indication to anesthetics or coelioscopy
* creatinine clearance less than 30 ml/min
* pregnant woman and protected persons
* no affiliation to social security
* unable to understand the information form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the reduction in morphine consumption | during the postoperative 48h

SECONDARY OUTCOMES:
Pain patient (ENS, total consumption of morphine) | during the hospitalization, to 10 days,1 month, 6 months and 12 months of surgery
quality of life (questionary SF-36) | 1 month, 6 month and 12 month of surgery
length of stay in hospital, percentage return home to 24 hours of surgery | to 24 hours of surgery
morbidity | during the study
resumption of work | after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Claude Tayar, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Chenevier-Mondor, Créteil, France